CLINICAL TRIAL: NCT00471341
Title: A Pilot Study to Determine the Effect of Celecoxib on Markers of Inflammation in Patients With Hypertension and Coronary Artery Disease
Brief Title: Effect of Celecoxib on Markers of Vascular Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 219-2001
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2007-05

CONDITIONS: Hypertension and Coronary Artery Disease
Keywords: arteriosclerosis; coronary disease; inflammation; COX-2 inhibition; hypertension
MeSH Terms: conditions — Hypertension; Coronary Artery Disease; Arteriosclerosis; Coronary Disease; Inflammation | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Celecoxib
Drug: placebo

SUMMARY:
This study involves a drug called celecoxib, which is commonly prescribed for people with arthritis. Arthritis is caused by inflammation of the joints or tissues. Inflammation also occurs in the blood vessels that lead to your heart, and the purpose of this study is to see if celecoxib can reduce the blood vessel inflammation associated with high cholesterol and heart disease.

DETAILED DESCRIPTION:
Chronic inflammation of the blood vessel wall is a hallmark of atherosclerosis. Elevated levels of low-density lipoprotein cholesterol (LDL-C), as well as blood pressure are known to be proinflammatory. Recent information suggests that acute ischemic events are associated with exacerbations in inflammation. Some data suggest that aspirin use is associated with suppression of markers of inflammation, and this response has been linked with improved outcome. Similarly, HMG Co-A Reductase inhibitors clearly reduce adverse outcomes in patients with atherosclerosis and recently, HMG Co-A Reductase inhibitor use has also been linked to reduction in inflammation. Due to the strong association of atherogenesis and plaque stability with inflammation, C-Reactive Protein (CRP), a marker of inflammation, has been evaluated as a potential tool for clinicians to assess cardiovascular risk, and has been found to be highly correlated. There is also evidence to suggest that cyclooxygenase 2 (COX-2) enzyme is expressed in plaque at regions which are vulnerable to rupture. Accordingly, this study is designed to investigate the potential reduction in vascular inflammation from a specific COX-2 inhibitor, celecoxib, as measured by a reduction from baseline of CRP, interleukin-6 (IL-6) and tumor necrosis factor - alpha (TNF-alpha). This is a double blind, placebo controlled pilot study in hypertensive patients with coronary artery disease and dyslipidemia, to evaluate the effect of celecoxib versus placebo on inflammatory markers. Patients will receive study drug for three months.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 50 years old
* Hypertension documented and treated according to the 6th report of the Joint National Committee on Detection and Evaluation of the treatment of high blood pressure (JNC VI)
* Documented coronary artery disease, defined as classic stable angina pectoris, previous myocardial infarction (more than 1 month ago) or unstable angina (more than 1 month ago), abnormal coronary angiogram, or concordant abnormalities on two different types of stress tests
* Dyslipidemia requiring medical therapy with HMG CoA Reductase inhibitors, and treated according to NCEP II guidelines for cholesterol lowering
* Diabetes, if treated according to ADA guidelines for diabetes
* Classic angina, if treated according to ACC/AHA guidelines for angina control
* Therapy with an HMG CoA Reductase inhibitor for at least 3 months
* Willingness to provide informed consent

Exclusion Criteria:

* PUD
* Coronary Artery Bypass Surgery or PTCA in the past 6 months
* Active infection
* Weight < 50Kg
* History of a hematologic bleeding disorder
* History of gastrointestinal bleeding
* Allergy to aspirin or celecoxib or other NSAIDs or sulfonamides
* Allergy or intolerance to HMG CoA Reductase inhibitor therapy
* Stroke within 1 month of enrollment
* History of a chronic inflammatory disease
* History of asthma
* History of hepatic disorder
* Advanced renal disease (Serum Creatinine > 3mg/dl)
* Anticipated need for therapy with NSAIDs within the 3 month period of the study
* Chronic therapy (14 consecutive days) with any NSAID in the last 30 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2002-07; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change in CRP

SECONDARY OUTCOMES:
Change in IL6
Change in TNF alpha
Change in BP
Change in indices of vascular function (FMD and vascular compliance)

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda M Cooper-DeHoff, Pharm D, Principal Investigator — University of Florida Faculty
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of Texas Health Science Center, Houston, Texas